CLINICAL TRIAL: NCT03769636
Title: Changes in Physical Activity in All Day Life (Steps, Distance, Periods, Max. Speed) in People With MS Before and After the Rehabilitation - A Prospective Observational Study
Brief Title: Changes in Physical Activity in All Day Life in People With MS Before and After Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, April Roger, Pricipal Investigator, Klinik Valens
Other Study IDs: BASEC Nr. 2017-00728
Record Dates: First submitted 2018-11-28; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Rehabilitation
Keywords: Multiple Sclerosis; In-patient rehabilitation; All day life activities; Walking capacity; Fatigue; Quality of life
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: GaitUp Physilog 5 — The primary outcomes are measured by the Physilog 5 (physical activity) at four different periods (T1-T4). Physilog 5 is worn for 4 weeks in total.
  The secondary outcomes are fatigue, measured by FSMC (fatigue scale for motor and cognitive functions questionnaire), self-rated health-related quality of life, measured by the EQ-5D (health-questionnaire) and self-rated walking capacity, measured by the MSWS-12 (Twelve Item MS Walking Scale).

SUMMARY:
The primary objective is to observe the impact of in-patient rehabilitation on physical activity in daily life using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.

The secondary objective is the association of changes in physical activity, self-rated walking capacity, self-rated fatigue and self-rated health-related quality of life, wich will be analysed for disease severity of the participants.

DETAILED DESCRIPTION:
Gait disorders are common in patients with multiple sclerosis (PwMS). Multidisciplinary in-patient rehabilitation conducted by specialized doctors, nurses and therapists can improve the ability to walk by tackling the problem with various approaches: by increasing strength in leg muscles, by improving balance, by increasing cardio- pulmonary fitness, by fitting walking aids, by reducing fatigue and cognitive deficits, by working out strategies to compensate for impairments, and by optimising medical treatment. The investigator's patients, who spend a lot of time (usually 2- 4 weeks) and effort for in-patient rehabilitation in Valens tell us, that this intensive therapy is usually effective and that their walking ability improves to a degree that is relevant in daily life. The scientific evidence for the effectiveness of in- patient rehabilitation is usually based on either clinical assessments of function (e.g. the 6 minute walking test) or on reports from PwMS, by using questionnaires e.g. about mobility or quality of life in daily life. Although clinical assessments provide important information about improvements of the functional capacity, they do not provide information about the impact of therapy on daily life. Patient reports, on the other hand, provide important information about the perceived impact in daily life, but the information is not objective. Objective information about the impact of rehabilitation on daily life is usually not available.

The primary objective therefore is to observe the impact of in-patient rehabilitation on physical activity in daily life using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.

The secondary objective is the association of changes in physical activity, self-rated walking capacity, self-rated fatigue and self-rated health-related quality of life, wich will be analysed for disease severity of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Planed rehabilitation in Valens between january 2018 and june 2019
* EDSS 2.0-6.5 (an EDSS 6.5 means the ability to walk 20 meters without resting, using constant bilateral assistance)
* German speaking
* Good function of upper limb, that the device can be fixed by participant himself
* Informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator plans to include 30 patients with multiple sclerosis with an EDSS 2.0-6.5, who come to Valens for rehabilitation between january 2018 and june 2019
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Changes in physical activity: Locomotion | Physical activity will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  The primary objective is to observe the impact of in-patient rehabilitation on physical activity in daily life in patients with MS (EDSS 2.0-6.5) using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.
  The following parameter represents the walking in daily life:
  - Locomotion: Percentage of locomotion (walking) per day The maximum value is 100%, the minumum value is 0%.
Changes in physical activity: Non-locomotion | Physical activity will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  The primary objective is to observe the impact of in-patient rehabilitation on physical activity in daily life in patients with MS (EDSS 2.0-6.5) using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.
  The following parameter represents the walking in daily life:
  - Non-locomotion: Percentage of non-locomotion (sitting, standing, lying) per day The maximum value is 100%, the minumum value is 0%.
Changes in physical activity: Level walking | Physical activity will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  The primary objective is to observe the impact of in-patient rehabilitation on physical activity in daily life in patients with MS (EDSS 2.0-6.5) using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.
  The following parameter represents the walking in daily life:
  - Level walking: Percentage of level walking per day The maximum value is 100%, the minumum value is 0%.
Changes in physical activity: Up walking | Physical activity will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  The primary objective is to observe the impact of in-patient rehabilitation on physical activity in daily life in patients with MS (EDSS 2.0-6.5) using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.
  The following parameter represents the walking in daily life:
  - Up walking: Percentage of up walking per day The maximum value is 100%, the minumum value is 0%.
Changes in physical activity: Down walking | Physical activity will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  The primary objective is to observe the impact of in-patient rehabilitation on physical activity in daily life in patients with MS (EDSS 2.0-6.5) using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.
  The following parameter represents the walking in daily life:
  - Down walking: Percentage of down walking per day The maximum value is 100%, the minumum value is 0%.
Changes in physical activity: Maximum steps | Physical activity will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  The primary objective is to observe the impact of in-patient rehabilitation on physical activity in daily life in patients with MS (EDSS 2.0-6.5) using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.
  The following parameter represents the walking in daily life:
  - Maximum steps: Maximal number of continuous steps in one walking bout (a walking bout is defined as walking more than two continuous steps).
  The maximum value is open, the minimum value is zero.
Changes in physical activity: Steps per hour | Physical activity will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  The primary objective is to observe the impact of in-patient rehabilitation on physical activity in daily life in patients with MS (EDSS 2.0-6.5) using miniature, wearable sensors, fixed on the shoes. These sensors record data about various aspects of walking. The information on the therapy effect on daily life can complement the clinical information and the patients' subjective report on therapy induced improvements.
  The following parameter represents the walking in daily life:
  - Steps per hour: Number of steps during all recorded walking bouts (the values are normalised per worn hours).
  The maximum value is open, the minimum value is zero.

SECONDARY OUTCOMES:
Changes in self-rated fatigue | Fatigue will first be measured 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  Fatigue will be measured by the Fatigue Scale for Motor and Cognitive Functions (FSMC). The FSMC is a 20-points-questionnaire with ten questions about cognitive fatigue and ten questions about motor fatigue. The questions are rated on a 5-point Likert-scale from 1 (does not apply at all) to 5 (applies completely). The total score ranges from a minimum of 20 points to a maximum of 100 points, sub-scores for cognitive and motor fatigue range from a minimum of 10 points to a maximum of 50 points. Higher scores indicate a higher perception of fatigue.
  The following comparisons are executed:
  * Comparison between T1 and T2
  * Comparison between T2 and T3
  * Comparison between T2 and T4
Changes in self-rated health-related quality of life: EQ-5D | Self-rated health-related quality of life will first be measured 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  Self-rated health will be measured by the questionnaire "health- related quality of life" (EQ-5D). The EQ-5D is a fife-points questionnaire about the topics "mobility", "self-care", "usual-activities", "pain/discomfort" and "anxiety/depression". The questions are rated with the following possibilities: "no problems", "some problems" and "extreme problems". On the basis of standardized calculations a index value is generated. The value ranges form zero to one. Higher values indicate a higher health-related quality of life.
  The following comparisons are executed:
  * Comparison between T1 and T2
  * Comparison between T2 and T3
  * Comparison between T2 and T4
Changes in self-rated walking capacity | Self-rated waking capacity will first be measured 4-6 weeks before rehabilitation (T1) in Valens, the week right before rehabilitation (T2), the week right after rehabilitation (T3) and 2 months after rehabilitation (T4).
  Self-rated walking capacity will be measured by the 12-Item MS Walking Scale (MSWS-12). The MSWS-12 is a twelve-points questionnaire to represent the impact of MS on walking capacity. The questions are rated on a five-point Likert-scale from 1 (not at all) to 5 (extremely). The total score ranges from a minimum of 12 points to a maximum of 60 points. Higher scores indicate a higher impact of MS on walking capacity.
  The following comparisons are executed:
  * Comparison between T1 and T2
  * Comparison between T2 and T3
  * Comparison between T2 and T4

OTHER OUTCOMES:
10 meter walking test (10TW) | 10TW will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the first week of rehabilitation (T2) and the third week of rehabilitation (T3).
  10TW will be assessed to see changes in walking speed.
Timed up and go (TUG) | TUG will first be assessed 4-6 weeks before rehabilitation (T1) in Valens, the first week of rehabilitation (T2) and the third week of rehabilitation (T4).
  TUG will be assessed to see changes in equilibrium and walking abilities.
2 minutes walking test (2MWT) | 2MWT will be assessed in the first week of rehabilitation (T2) and in the third week of rehabilitation (T3).
  2MWT will be assessed to see changes in walking speed and distance
Stair measure test (ST) | ST will be assessed in the first week of rehabilitation (T2) and in the third week of rehabilitation (T3).
  ST will be assessed to see changes in speed and walking abilities on stairs.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Valens, Valens, St.Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heesen C, Bohm J, Reich C, Kasper J, Goebel M, Gold SM. Patient perception of bodily functions in multiple sclerosis: gait and visual function are the most valuable. Mult Scler. 2008 Aug;14(7):988-91. doi: 10.1177/1352458508088916. Epub 2008 May 27. PMID 18505775
- [Background] Campbell E, Coulter EH, Mattison PG, Miller L, McFadyen A, Paul L. Physiotherapy Rehabilitation for People With Progressive Multiple Sclerosis: A Systematic Review. Arch Phys Med Rehabil. 2016 Jan;97(1):141-51.e3. doi: 10.1016/j.apmr.2015.07.022. Epub 2015 Aug 14. PMID 26281954
- [Background] Khan F, Amatya B. Rehabilitation in Multiple Sclerosis: A Systematic Review of Systematic Reviews. Arch Phys Med Rehabil. 2017 Feb;98(2):353-367. doi: 10.1016/j.apmr.2016.04.016. Epub 2016 May 20. PMID 27216225
- [Background] Beer S, Khan F, Kesselring J. Rehabilitation interventions in multiple sclerosis: an overview. J Neurol. 2012 Sep;259(9):1994-2008. doi: 10.1007/s00415-012-6577-4. Epub 2012 Jul 8. PMID 22772357
- [Background] Gunn H, Markevics S, Haas B, Marsden J, Freeman J. Systematic Review: The Effectiveness of Interventions to Reduce Falls and Improve Balance in Adults With Multiple Sclerosis. Arch Phys Med Rehabil. 2015 Oct;96(10):1898-912. doi: 10.1016/j.apmr.2015.05.018. Epub 2015 Jun 10. PMID 26070975
- [Background] Stevens V, Goodman K, Rough K, Kraft GH. Gait impairment and optimizing mobility in multiple sclerosis. Phys Med Rehabil Clin N Am. 2013 Nov;24(4):573-92. doi: 10.1016/j.pmr.2013.07.002. Epub 2013 Sep 7. PMID 24314677
- [Background] Schwartz CE, Ayandeh A, Motl RW. Investigating the minimal important difference in ambulation in multiple sclerosis: a disconnect between performance-based and patient-reported outcomes? J Neurol Sci. 2014 Dec 15;347(1-2):268-74. doi: 10.1016/j.jns.2014.10.021. Epub 2014 Oct 18. PMID 25455299
- [Background] Fjeldstad C, Fjeldstad AS, Pardo G. Use of Accelerometers to Measure Real-Life Physical Activity in Ambulatory Individuals with Multiple Sclerosis: A Pilot Study. Int J MS Care. 2015 Sep-Oct;17(5):215-20. doi: 10.7224/1537-2073.2014-037. PMID 26472942
- [Background] Casey B, Coote S, Donnelly A. Objective physical activity measurement in people with multiple sclerosis: a review of the literature. Disabil Rehabil Assist Technol. 2018 Feb;13(2):124-131. doi: 10.1080/17483107.2017.1297859. Epub 2017 Mar 13. PMID 28285547